CLINICAL TRIAL: NCT03209115
Title: Influence of Calcium Hydroxide Chlorhexidine Combination vs. Calcium Hydroxide as an Intra Canal Medicamentson Postoperative Flare -up Following Two-Visit Endodontic Retreatment Cases
Brief Title: Influence of Calcium Hydroxide Chlorhexidine Combination vs. Calcium Hydroxide as an Intra Canal Medicaments in Retreatment Cases
Acronym: med
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hind Midhat AbdulGader Hussein, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hind
Record Dates: First submitted 2017-07-03; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Postoperative Flare up
MeSH Terms: interventions — Chlorhexidine; Calcium Hydroxide

STUDY DESIGN:
Intervention Model Description: Intracanal medication
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- calcium hydroxide and chlorhexidine (Active Comparator): Removal of old root canal filling and placing calcium hydroxide and chlorehexidine as intracanal medication
  Interventions: Drug: combination of calcium hydroxide and chlorhexidine
- calcium hydroxide (Active Comparator): Removal of old root canal filling and placing calcium hydroxide as intracanal medication
  Interventions: Drug: Calcium Hydroxide

INTERVENTIONS:
Drug: combination of calcium hydroxide and chlorhexidine — placement of calcium hydroxide and chlorhexidine as intracanal medicament after removal of old filling and mechanical preparation of root canal
  Arms: calcium hydroxide and chlorhexidine
Drug: Calcium Hydroxide — placement of calcium hydroxide as intracanal medicament after removal of old filling and mechanical preparation of root canal
  Arms: calcium hydroxide

SUMMARY:
Influence of Calcium hydroxide Chlorhexidine Combination vs. Calcium Hydroxide as an Intra canal Medicamentson Postoperative flare -up following two-Visit Endodontic Retreatment cases

DETAILED DESCRIPTION:
1. Each patient will be anesthetized with the same solution, 40 mg articaine hydrochloride + 0.006 mg/mL epinephrine hydrochloride (Ultracaine DS; Aventis Pharma, Istanbul, Turkey).
2. The standard procedure for each group at the first appointment included rubber dam isolation,removing of previous coronal restorations, and root canal filling materials. The removal of previous root canal fillings will be performed with one of these: Gates Glidden drills, hand files, heated pluggers, and Ni-Ti rotary instruments.
3. After the removal of previous root canal fillings, the working lengths were determined by apex locator and periapical radiographs 1 mm from the apexes.
4. Chemo-mechanical preparation of root canals will be made with the master apical files ranged from #25 to #70 depending on the initial diameter or preparation of the root canals.

   Irrigation was performed with 2.5% NaOCl after each instrument in all cases. At the end of instrumentation, the final irrigation was made by saline, and the root canals were dried with paper points.
5. In the 1st group the root canals will be medicated with a calcium hydroxide paste for 7 days.(calcium hydroxide injectable paste Metapex , 2.2g paste in a 1 syringe).

   In the 2nd group the root canals will be medicated with a calcium hydroxidechlorhexidine paste for 7 days. The paste consists of 1.2 g Ca(OH)2 powder per 1 mL 0.2% chlorhexidine in water. The teeth in both groups will be closed with a sterile dry cotton pellet and a minimum of 3 mm of temporary restorative material.
6. In the next appointment, the tooth was reopened, the intra-canal paste will be removed and a patency file (size 08 Flexofile; Dentsply-Maillefer) was pushed through the foramen.

Master apical file will be checked again and then master cones will be placed and radiographed. Obturation will be done using lateral compaction technique with AD seal resin sealer using spreader for placement of auxiliary cones.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' needs retreatment.
2. Patients in good health with no systemic disease (American Society of Anesthesiologists Class II)
3. Age range is between 20 and 50 years.
4. Patients who can understand the categorical tool (points)for measurement
5. Patients able to sign informed consent.

Exclusion Criteria:

1. Complicating systemic disease
2. Having severe pain and/or acute apical abscesses
3. Being under 18 years of age
4. Using antibiotics or corticosteroids

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2017-07-08 (Estimated); Primary Completion 2017-09-08 (Estimated); Study Completion 2018-07-08 (Estimated)

PRIMARY OUTCOMES:
Postoperative flare up (pain and swelling ) will be measured as below after 7 days from first visit postoperative pain | 7 days
  categorical ( 4 points)
  1. no pain
  2. Mild pain: recognizable but not discomforting pain that required no analgesics.
  3. Moderate pain: discomforting but bearable pain(analgesics if used were effective in relieving pain)
  4. Severe pain: difficult to bear (analgesics were effective in relieving pain). Patients with severe postoperative pain and/or occurrence of swelling were classified as flare-ups.3 Objectively : percussion test

CONTACTS AND LOCATIONS:
Overall Officials: Geraldine M Ahmed, Assistant professor, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No